CLINICAL TRIAL: NCT01821755
Title: Development, Implementation and Evaluation of a Foster Parent Intervention
Brief Title: Effectiveness of a Foster Parent Intervention: Results of a Trial
Acronym: PVO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Femke vanschoonlandt, PhD Student, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID0032
Record Dates: First submitted 2013-02-19; First posted 2013-04-01 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Problematic Behavior in Children; Parent-child Problem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral: Foster parent intervention (Experimental): Foster parents receive a foster parent intervention consisting of 10 individual home visits and three group sessions. Duration of the intervention is four months
  Interventions: Behavioral: Foster parent intervention
- Control (No Intervention): waiting-list control group who receive care-as-usual

INTERVENTIONS:
Behavioral: Foster parent intervention — parent management training for foster parents, consisting of 10 individual home visits and 3 group sessions. Duration is four months
  Arms: Behavioral: Foster parent intervention

SUMMARY:
The hypothesis of the study is that the intervention leads to a reduction in foster children's externalizing problems and foster parents' parenting stress and that this in turn leads to a reduction in the number of breakdowns of foster placements.

ELIGIBILITY:
Inclusion Criteria:

* foster child has a borderline or clinical score on one of the small-band externalizing scales or the broad-band externalizing scale of the Child Behavior Checklist (CBCL)

Exclusion Criteria:

foster child:

* has a mental retardation,
* autism,
* uses psychotropic medication in an inconsistent way,
* behavioral problems are the result of medical problems or medication, foster parents:
* have insufficient knowledge of Dutch,
* have low cognitive abilities,
* are already receiving professional support for the foster child's externalizing problems,
* are divorcing.

Moreover, foster placements were excluded if at least two of the following criteria were present:

* foster parents considered terminating the foster placement during the past two months
* were experiencing psychological distress (measured with the General Health Questionnaire (GHQ; Koeter & Ormel, 1991) and defined as a score ≥ 2),
* their foster child had a sum score above 3 (for children < 6 years) or 5 (for children ≥ 6 years) on the critical CBCL-items.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Change in foster child's externalizing problems from baseline to post-intervention (3.5 months later) | Assessed at two time points: at baseline (before the start of the intervention) en post-intervention (immediately after the intervention has ended, which is on average 3.5 months after the baseline measurement)
  T-score for the externalizing subscale of the Child Behavior Checklist (CBCL)
Change in foster child's externalizing problems from post-intervention to follow-up (3 months later) | Assessed at post-interventio (immediately after the intervention has ended, which is about 3.5 months after the baseline measurement) and at follow-up (which is thee months later than the post-intervention measurement).
  The T-score of the Externalizing scale of the Child Behavior Checklist (CBCL)

SECONDARY OUTCOMES:
Change in foster parent's parenting stress from baseline to post-intervention (3.5 months later) | Assessed at two time points: at baseline (before the start of the intervention) en post-intervention (immediately after the intervention has ended, which is on average 3.5 months after the baseline measurement)
  Nijmegen Questionnaire for the Parenting Situation
Change in foster mother's parenting stress from post-intervention to follow-up (3 months later) | Assessed at post-interventio (immediately after the intervention has ended, which is about 3.5 months after the baseline measurement) and at follow-up (which is thee months later than the post-intervention measurement).
  The Nijmegen Questionnaire for the parenting situation
Client satisfaction | At post-intervention (immediately after the intervention has ended, which is on average 3.5 months later than the baseline measurment
  Dutch Questionaire for client satisfaction and effect
Change in foster mother's parenting behavior from baseline to post-intervention (3.5 months later) | Assessed at two time points: at baseline (before the start of the intervention) en post-intervention (immediately after the intervention has ended, which is on average 3.5 months after the baseline measurement)
  The Ghent Parenting Behavior Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Brussels, Vlaams-Brabant, Belgium